CLINICAL TRIAL: NCT05723315
Title: Effect of rhBNP on Coronary Microcirculation in Patients With Acute ST-segment Elevation Myocardial Infarction After Primary PCI
Brief Title: Effect of rhBNP on CMD in Patients With STEMI After PPCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HenanICE202301
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group 1 (Experimental): The experimental group was given neoptin within 3h after PCI for 72 hours (first at 1.5μg /kg intravenous load, then at 0.015μg /kg/min).
  Interventions: Drug: recombinant human B-type natriuretic peptide
- Control Gruop (No Intervention): The experimental group was given an intravenous infusion of the same amount of normal saline

INTERVENTIONS:
Drug: recombinant human B-type natriuretic peptide — The recombinant human B-type natriuretic peptide produces physiological effects by imitating endogenous B-type natriuretic peptide
  Other Names: rhBNP
  Arms: Experimental Group 1

SUMMARY:
The target population of this interventional study was STEMI patients. Primary discussion: Early rhBNP reduces microcirculation obstruction in STEMI patients undergoing primary PCI

DETAILED DESCRIPTION:
Direct percutaneous coronary intervention is the preferred reperfusion strategy for acute ST-segment elevation myocardial infarction. During the opening of infarct-related vessels, 5%-50% of patients showed slow flow or no reflow and other coronary microcirculation dysfunction, which aggravated myocardial injury and increased the incidence and mortality of heart failure. Studies have shown that recombinant human brain natriuretic peptide (rhBNP) can reduce reperfusion injury and reduce myocardial infarction area CMD. Prolonged ischemia leads to rapid depletion of intracellular ATP and tissue metabolic acidosis. Blood flow irrigation during reperfusion leads to decreased levels of ATP precursors, calcium overload in mitochondria, release of a large number of inflammatory factors and oxygen free radicals, which can lead to injury or death of myocardial and endothelial cells. rhBNP can enhance the activity of antioxidant enzymes, reduce the irreversible oxidative damage caused by free radicals to myocardium, reduce the myocardial infarction area during ischemia reperfusion, and may reduce the reperfusion injury and protect the viable myocardium.

ELIGIBILITY:
Inclusion Criteria:

* STEMI
* PPCI within 24 hours of symptom onset
* Target vessel QFR-MR>250mm Hg*s/m

Exclusion Criteria:

* claustrophobia
* Postoperative TIMI grade 0-1
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
MVO/LV(%) | 3-14 days after PPCI
  Microvascular obstruction assessed by magnetic resonance imaging

SECONDARY OUTCOMES:
LGE/LV(%) | 3-14 days and 90±7 days after PPCI
  Cardiac magnetic resonance imaging
IMH | 3-14 days after PPCI
  Intramuscular hemorrhageCardiac assessed by magnetic resonance imaging
MVO/LV(%) | 30±7 days after PPCI
  Microvascular obstruction assessed by magnetic resonance imaging
LVEDV(ml) | 3-14 days and 90±7 days after PPCI
  Assessed by magnetic resonance imaging
LVESV(ml) | 3-14 days and 90±7 days after PPCI
  Assessed by magnetic resonance imaging
Troponin (highest value) | 3-14 days after PPCI
  Troponin (highest value)
MACCEs | 7days，30days，3months，6 months
  Major Adverse Cardiac and Cerebrovascular event：Death, nonfatal myocardial infarction, heart failure, revascularization, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, MD, Study Chair — Fuwai central China cardiovascular hospotial

IPD SHARING:
Plan to Share IPD: No